CLINICAL TRIAL: NCT02689609
Title: Dosimetric Predictors of Hypothyroidism After Radical Intensity-modulated Radiation Therapy for Non-metastatic Nasopharyngeal Carcinoma
Brief Title: Post-radiation Hypothyroidism After IMRT for Nasopharyngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: City University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Victor H.F. Lee, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: Version 1.0
Record Dates: First submitted 2016-02-15; First posted 2016-02-24 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Hypothyroidism; Complications
Keywords: Nasopharyngeal carcinoma; Intensity-modulated radiation therapy; Hypothyroidism; Predictors
MeSH Terms: conditions — Hypothyroidism; Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single arm: All patients will receive intensity-modulated radiation therapy (IMRT) with or without adjunct chemotherapy as standard of care. They will have baseline pre-treatment and post-IMRT serum thyroid function test at least yearly after IMRT.
  Interventions: Radiation: Intensity-modulated radiation therapy

INTERVENTIONS:
Radiation: Intensity-modulated radiation therapy — All patients will receive intensity-modulated radiation therapy with or without chemotherapy as usual standard of care in our institution.

SUMMARY:
The investigators evaluate if there are radiation dosimetric parameters for the prediction of biochemical and clinical hypothyroidism after intensity-modulated radiation therapy (IMRT) for non-metastatic nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
Eligible patients include those with previously untreated non-metastatic nasopharyngeal carcinoma (NPC) who will receive only one course of radical IMRT with or without adjunct chemotherapy for their NPC as curative treatment. Patients who have a history of any thyroid disorders, pituitary disorders, prior thyroid surgery or a drug history of thyroxine (T4) or triiodothyronine (T3) are excluded. Patients who have a history of radiation therapy to other areas are also excluded. Pretreatment investigations and workup include serum hematology, biochemistry, antibodies against Epstein-Barr virus (EBV) viral capsid antigen (VCA) and early antigen (EA), fabrication of customized head and neck thermoplastic cast for subsequent contrast-enhanced computed tomography (CT) scan of the head and neck region down to mid-thoracic region in IMRT treatment position with 3mm thickness, as well as T1-sequence, T2-sequence and gadolinium-enhanced magnetic resonance imaging (MRI) of the head and neck region by a 3-tesla scanner with the images co-registered with the planning head and neck CT images for detailed target and organ-at-risk (OAR) delineation and IMRT planning. A separate contrast-enhanced CT scan of the thorax and abdomen will also be performed to rule out distant metastasis.

The gross tumour volumes of both the primary tumour (GTV-P) and the radiologically involved cervical nodes (GTV-N) are outlined on the planning CT images with the aid of co-registered MRI images. Subsequently clinical target volume (CTV-70) and planning target volume containing CTV-70 with a 3mm margin (PTV-70) are generated to take into account the microscopic disease spread, physiological body motions and set-up errors respectively. Another CTV-66 encompassing the high risk areas including the posterior half of the maxillary sinuses, nasal cavities, parapharyngeal spaces, styloid processes, basi-occiput, basi-sphenoid, clivus, foramina rotunda and ovale, pterygopalatine fossae, pterygomaxillary fissures, infra-orbital fissures, cavernous sinuses and level Ib and level V nodal stations is also contoured. A corresponding PTV-66 with a 3mm margin encompassing CTV-66 is created by boolean operations of the treatment planning system which is also used for IMRT optimization and planning. All OARs including brainstem, spinal cord, globes, optic nerves, optic chiasm, lenses, temporomandibular joints, temporal lobes, auditory nerves, cochleae, mandible, oral cavity, larynx, parotid glands, vestibules, pituitary and thyroid are to be contoured manually. During IMRT optimization, the maximum dose of brainstem, optic nerves and chiasm must be <=54 Gy (allowing 0.1cc brainstem <60 Gy) and spinal cord <=45 Gy (allowing 0.1cc spinal cord <48 Gy). Efforts will also made to limit mean dose of parotid glands to 26 Gy whenever possible and dose to the lenses and temporal lobes as low as reasonably achieved without compromising dose coverage to the PTVs. No dose constraint is to be given to the thyroid and pituitary during optimization of all IMRT plans.

A 7 to 9 field IMRT plan delivered by step-and-shoot technique with a 6-megavoltage linear accelerator will be generated by Eclipse Treatment Planning System. A total dose of 70 Gy and 66 Gy was prescribed to PTV-70 and PTV-66 respectively, all in 33 to 35 fractions over 6.5 to 7 weeks by simultaneous accelerated radiation therapy technique (SMART). The whole neck was irradiated with IMRT and no matching anterior field to the lower neck was noted. This has been the standard prescription and practice in our institution for the past 10 years. Positional verification with on-board imaging was performed before IMRT commencement. It was repeated again daily immediately before the first 3 fractions of IMRT and then weekly afterwards during the whole course of IMRT, to track any anteroposterior and lateral body displacements.

All patients had routine 6-site nasopharyngeal biopsies at 8 weeks after IMRT to confirm local clinical remission. Repeated nasopharyngeal biopsies were performed at 10 weeks and 12 weeks after IMRT if residual tumour cells were still observed in previous post-IMRT nasopharyngeal biopsies. Additional radiation therapy in the form of intracavitary brachytherapy, stereotactic radiation therapy or IMRT would be given if patients developed local persistence at 12 weeks after IMRT. For patients confirmed to be local clinical remission, they received regular clinical follow up and imaging surveillance every 3 to 4 months for the 1st year after IMRT, then every 4 to 6 months for the 2nd and 3rd year and yearly afterwards to monitor for any treatment-related chronic complications and relapse. Blood tests for thyroid function tests including free T4 and thyroid stimulating hormone (TSH) will be arranged at least once yearly to monitor post-IMRT hypothyroidism. Biochemical hypothyroidism is defined as either elevation of TSH above the upper normal limit or reduced free T4 below the lower normal limit or both, without the presence of clinical symptoms of hypothyroidism. Clinical hypothyroidism is defined as the presence of biochemical abnormalities of thyroid function same as that defined for biochemical hypothyroidism together with the presence of clinical symptoms of hypothyroidism. Those who are found to have clinical hypothyroidism will receive thyroxine supplement starting with 50 micrograms daily with repeated serum thyroid function tests 2 to 3 months later followed by dose titration if necessary, then every 6 to 12 months thereafter when therapeutic dosage was reached.

Univariable and multivariable binary logistic regression will be performed for dosimetric predictors of biochemical and clinical hypothyroidism. All statistical analyses will be performed by Statistical Package for Social Sciences (SPSS) and statistical significance is defined as p-value <0.05 (two-sided).

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated non-metastatic NPC who are planned to receive radical intensity-modulated radiation therapy with or without adjunct chemotherapy.

Exclusion Criteria:

* Patients who are not able to give written informed consent
* Patients who are pregnant or lactating at the time of written consent
* Patients who have significant cardiovascular, cerebrovascular and psychiatric illness as judged serious by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients included those with previously untreated non-metastatic nasopharyngeal carcinoma (NPC) who received only one course of radical IMRT with or without adjunct chemotherapy for their NPC as curative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Biochemical hypothyroidism | Through study completion, an average of 3 years
  Time from IMRT to development of biochemical hypothyroidism

SECONDARY OUTCOMES:
Clinical hypothyroidism | Through study completion, an average of 3 years
  Time from IMRT to development of clinical hypothyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Victor HF Lee, MD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.